CLINICAL TRIAL: NCT05649280
Title: Safety Evaluation of DREPADOM - Home Care Services and Hospitalizations for Sickle Cell Disease Patients
Acronym: DREPADOM
Status: Completed | Type: Observational
Sponsor: Soutien aux Actions contre les Maladies du Globule Rouge (Other)
Responsible Party: Sponsor
Other Study IDs: AIR LIQUIDE HEALTH CARE
Record Dates: First submitted 2022-06-01; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to evaluate the incidence of ACS within the DREPADOM system and compare it to expected incidences of ACS (historic cohorts of PRESEV1 and PRESEV2)

DETAILED DESCRIPTION:
This prospective, observational study will take place, as follows:

Calculation of the PRESEV score in the ER will determine or not eligibility of the patient in the DREPADOM structure. With a low score, a patient is eligible for home monitoring and after duly provided information, can sign a patient consent for the use of personal medical data.

The coordinating nurse from DREPADOM can then set up a whole network, with the delivery of oxygen supply at the patient's house, dispatch of a medical prescription to a neighboring pharmacy and daily visits from homecare service providers. Both opioids and parenteral hydration and treatments can be prescribed and daily visits, up to three, are programmed. As such, the patient receives a minimum of 1 visit per day from a nurse for monitoring and is provided with a medical oxygen concentrator for home use (3L/min continuously or for at least 15h/day) and parenteral hydration. In addition, patients are called daily by general practitioners or SCD experts, for teleconsultations.

The DREPADOM coordinating nurse is in constant interaction with nurses/providers of homecare services/medical doctors and status and evolution of the patient's global condition is reported both through the constant contact with the coordinating nurse from DREPADOM and in a dedicated software (Link4Life), with monitoring of blood pressure, temperature, respiratory rate, pain, etc… Link4Life is a software tool developed especially for home monitoring. It is adaptable to specific disorders, fully complies with the French Law for Health Data management and allows data extraction. Link4Life has been adapted to SCD in full collaboration with SCD medical experts of the Henri Mondor hospital. It is to be noted that all medical doctors (general practitioners or SCD experts), as well as coordinating and visiting nurses have all access to this application. As such, Link4Life will gather and capture all patient data.

When reporting patients' clinical parameters daily in the dedicated app (controlled by the DREPADOM team of experts), alerts are generated in the software when these are above or below determined thresholds. The medical team of experts from DREPADOM then takes over for daily teleconsultations and medical decisions for pursuing home monitoring or hospital admittance.

Of important note, a patient can be included twice in the DREPADOM study, for two distinct VOCs. Indeed, the PRESEV1 study highlighted that each crisis is unique and should be treated accordingly.

Data capture will be done through the Link4Life software, as well as extraction for data analysis.

* Open-label
* Blind
* Number of treatment arms:

Single arm

Multi arms specify the number of arms:

* Not Controlled
* Controlled, specify the comparator:

Versus placebo Versus reference product Versus other (specify) -Randomized: Parallel group Cross over Other (specify)

-Intervention (gas and/or drug, and/or device, and/or service /study arm):

ELIGIBILITY:
Inclusion Criteria:

* SS or Sβ0
* Adult patients with a low PRESEV score

Exclusion Criteria:

* SC/Sβ+ patients
* SCD adult patients with an intermediate or high PRESEV score
* Pregnant or breastfeeding women
* Homeless patient
* Patients without Social Security
* Patient deprived of liberty by judicial or administrative decision or patient under guardianship

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sickle Cell Disease (SCD) is the most widespread genetic disease in the world. With an incidence rate of approximately 1/3000 newborns each year in France, International Standards consider SCD a rare disease. However, in the Ile-de-France region, that incidence drops to 1/435 newborns, rendering SCD a major territorial issue. It is estimated that more than 10 000 SCD patients live in this region, which represents approximately 30% of the French SCD population and 10% of the European SCD population.
  Vaso-occlusive crisis (VOC) or acute bone pain vaso-occlusion is a characteristic manifestation of SCD and represents the first cause of patients 'hospitalizations. Moreover, 16% of VOCs can develop into a potentially severe complication: the acute chest syndrome (ACS).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of acute chest pain | 30 months
  The primary endpoint is the incidence of Acute chest pain complications developed by patients in the DREPADOM system ( Home Care Services and Hospitalizations for Sickle Cell Disease Patients) and comparison with the historical cohorts of( PRESEV1 and PRESEV2 studies).

SECONDARY OUTCOMES:
Incidence of clinical complications associated to Sickle cell disease | 30 months
  * Transfusions and comparison with historical cohorts of PRESEV1 and PRESEV2 studies
  * Patient admission in intensive care unit and comparison with historical cohorts of PRESEV1 and PRESEV2 studies
  * Mortality and comparison with historical cohorts of PRESEV1 and PRESEV2 studies

CONTACTS AND LOCATIONS:
Overall Officials: Pablo BARTOLUCCI, PROFESSOR, Principal Investigator — Soutien aux Actions contre les Maladies du Globule Rouge
Locations (1):
- Henri Mondor Hospital, Créteil, France